CLINICAL TRIAL: NCT04140396
Title: A Prospective Comparison of Continuous Intravenous Lidocaine Infusion Versus Placebo for Rib Fracture Analgesia
Brief Title: Continuous Intravenous Lidocaine Infusion Versus Placebo for Rib Fracture Analgesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of personnel and lack of funding for the study drug
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 53087
Record Dates: First submitted 2019-10-16; First posted 2019-10-25 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Comparator (Placebo Comparator): Participants will receive placebo infusion consisting of normal saline
  Interventions: Drug: Saline infusion
- Active Comparator (Active Comparator): Participants will receive a lidocaine infusion
  Interventions: Drug: Lidocaine infusion

INTERVENTIONS:
Drug: Saline infusion — Normal saline infusion at 10mL/hour
  Arms: Placebo Comparator
Drug: Lidocaine infusion — Lidocaine infusion at 1.0mg/kg/hr
  Arms: Active Comparator

SUMMARY:
The current cornerstone of pain control for rib fractures is oral and intravenous opioids, especially in the form of patient-controlled analgesia (IV PCA), which are are associated with multiple adverse effects including sedation, respiratory depression, cough suppression, and increased risk of delirium.

In the past few decades, intravenous lidocaine infusion (IVL) has emerged as a new tool in the arsenal of multimodal analgesia. Multiple randomized clinical trials have indicated that IVL is overall well tolerated and have shown other beneficial effects such as anti-inflammatory properties. To this date, there have been no published randomized clinical trials (RCT) evaluating the effectiveness of IVL in management of traumatic rib fracture pain.

Therefore, the purpose of this study is to evaluate whether IV Lidocaine infusion can provide improved pain control as demonstrated by decreased OME consumption at 24 and 48 hours compared to placebo in adult patients with acute traumatic rib fractures.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients admitted to Stanford Health Care with two or more acute traumatic rib fractures

Exclusion Criteria:

* hemodynamically instability
* mechanical ventilation
* polytrauma (defined as bone or organ injury outside the thorax)
* pregnancy
* incarceration
* local anesthetic allergy or contraindications to lidocaine (Stokes-Adams syndrome, Wolff-Parkinson-White syndrome, or severe degrees of sinoatrial, atrioventricular, or intraventricular block)
* chronic opioid use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Healthcare, Stanford, California, United States

REFERENCES:
- [Background] Hollmann MW, Durieux ME. Local anesthetics and the inflammatory response: a new therapeutic indication? Anesthesiology. 2000 Sep;93(3):858-75. doi: 10.1097/00000542-200009000-00038. No abstract available. PMID 10969322
- [Background] Flagel BT, Luchette FA, Reed RL, Esposito TJ, Davis KA, Santaniello JM, Gamelli RL. Half-a-dozen ribs: the breakpoint for mortality. Surgery. 2005 Oct;138(4):717-23; discussion 723-5. doi: 10.1016/j.surg.2005.07.022. PMID 16269301
- [Background] Gordy S, Fabricant L, Ham B, Mullins R, Mayberry J. The contribution of rib fractures to chronic pain and disability. Am J Surg. 2014 May;207(5):659-62; discussion 662-3. doi: 10.1016/j.amjsurg.2013.12.012. Epub 2014 Jan 31. PMID 24612969
- [Background] Battle CE, Hutchings H, Evans PA. Risk factors that predict mortality in patients with blunt chest wall trauma: a systematic review and meta-analysis. Injury. 2012 Jan;43(1):8-17. doi: 10.1016/j.injury.2011.01.004. Epub 2011 Jan 22. PMID 21256488

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: Participants will receive a lidocaine infusion at 1.0mg/kg/hr.
Period: Overall Study
Arm/Group | Placebo Comparator | Active Comparator
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active Comparator
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Oral Morphine Milligram Equivalent (OME) Consumption at 24 Hours
Description: MME = morphine milligram equivalent
Time Frame: After 24 hours of treatment
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Active Comparator
Number analyzed (Participants) | 1
MME | 7.5 (NA) — Standard deviation not calculable for n of 1

2. Secondary Outcome: Cumulative Oral Morphine Milligram Equivalent (OME) Consumption at 48 Hrs
Time Frame: After 48 hours of treatment
Population: No data were collected for this outcome, patient was discharged prior to this time point.
Arm/Group | Active Comparator
Number analyzed (Participants) | 0

3. Secondary Outcome: Pain Score
Description: Pain scores at rest rated using the Numeric Rating Scale (NRS) of 0-10, where 0 is no pain and 10 is the worst imaginable
Time Frame: Baseline and 1, 10, 13, 16, and 17 hours post-lidocaine infusion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator
Number analyzed (Participants) | 1
score on a scale
  Pre-infusion baseline | 1 (NA) — Standard deviation not calculable for n of 1
  1 hour post-infusion | 1 (NA) — Standard deviation not calculable for n of 1
  10 hours post-infusion | 0 (NA) — Standard deviation not calculable for n of 1
  13 hours post-infusion | 0 (NA) — Standard deviation not calculable for n of 1
  16 hours post-infusion | 4 (NA) — Standard deviation not calculable for n of 1
  17 hours post-infusion | 2 (NA) — Standard deviation not calculable for n of 1

4. Secondary Outcome: Incentive Spirometry Volumes
Description: An incentive spirometer is a device that measures how deeply you can inhale. Higher volumes indicate greater ability to inhale.
Time Frame: Pre-infusion baseline and 24 hours post-infusion
Population: Standard deviation not calculable for n of 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Active Comparator
Number analyzed (Participants) | 1
mL
  Pre-infusion baseline | 1500 (NA) — Standard deviation not calculable for n of 1
  24 hours post-infusion | 1500 (NA) — Standard deviation not calculable for n of 1

5. Secondary Outcome: PIC Score
Description: PIC score is a composite score comprising pain level, ISV, and cough strength. PIC scores range from 1-10 with one being severe pain, inability to perform incentive spirometry, and absent cough and 10 being controlled pain, an incentive spirometry volume above goal volume (set by respiratory therapist), and strong cough.
Time Frame: Time 0, 24 hours, 48 hour, and 72 hours.
Population: Data were not collected for this outcome measure.
Arm/Group | Active Comparator
Number analyzed (Participants) | 0

6. Secondary Outcome: Length of Hospital Stay
Description: Number of hours stayed at the hospital from the day of operation till the day of discharge.
Time Frame: 29 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Active Comparator
Number analyzed (Participants) | 1
hours | 29 (NA) — Standard deviation not calculable for n of 1

7. Secondary Outcome: Inflammatory Biomarkers
Description: Proinflammatory markers (IL6, IL8, IL-1β, TNF-α) and f anti-inflammatory markers (IL10)
Time Frame: Time 0, 24 hours, and 48 hour
Population: Data were not collected for this outcome measure.
Arm/Group | Active Comparator
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Pulmonary Complication Events
Description: Pulmonary complications include ARDS, pneumonia, aspiration, empyema, etc.
Time Frame: 29 hours
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Active Comparator
Number analyzed (Participants) | 1
events | 0 (NA) — Standard deviation not calculable for n of 1

ADVERSE EVENTS:
Time Frame: 29 hours
Arm/Group | Active Comparator
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
This study did not meet its planned enrollment size and did not achieve statistical significance as prespecified in the study protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT04140396/Prot_SAP_000.pdf